CLINICAL TRIAL: NCT03382119
Title: Increased Liver Stiffness: A Study of Acoustic Radiation Force Impulse (ARFI) Elastography
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Frank DiPaola, Assistant Professor, University of Michigan
Other Study IDs: HUM 130099
Record Dates: First submitted 2017-12-13; First posted 2017-12-22 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Liver Fibroses
Keywords: liver stiffness Fontan
MeSH Terms: conditions — Liver Cirrhosis | interventions — Ultrasonography; Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients having Fontan cardiac surgery: This group includes pediatric patients, aged 2-5 years, who have had a Fontan operation. This surgery corrects a heart defect found at birth in which the heart has only one ventricle.
  Patients will have an Ultrasound with ARFI imaging.
  Interventions: Device: Ultrasound with ARFI (acoustic radiation force impulse); Device: Ultrasound with backscatter imaging
- Patients with Liver disease: This group includes pediatric patients, aged 2-5 years, who have chronic liver disease caused by biliary atresia.
  Patients will have an Ultrasound with ARFI imaging.
  Interventions: Device: Ultrasound with ARFI (acoustic radiation force impulse); Device: Ultrasound with backscatter imaging

INTERVENTIONS:
Device: Ultrasound with ARFI (acoustic radiation force impulse) — This technology uses sound waves to measure the stiffness of tissue.
  Other Names: elastography
Device: Ultrasound with backscatter imaging — This ultrasound tool gathers data from the waves returning from imaged tissue.

SUMMARY:
The goal of this study is to determine if ultrasound tools can be used to detect liver stiffness. Acoustic radiation force impulse (ARFI) elastography and backscatter will be used to see if they can detect liver stiffness in different populations of patients with liver disease.

The study is measuring liver stiffness in pediatric patients aged 2-5 years. Patients either have had a Fontan cardiac surgery or have liver disease.

Ultrasound scanning takes images of the liver and has much lower risks for patients. ARFI elastography and other tools can be used to measure liver stiffness.

DETAILED DESCRIPTION:
If patients have liver congestion, reversing it could prevent liver fibrosis, which cannot be treated. Liver fibrosis has serious health risks and is associated with a higher chance of developing liver cancer later in life.

Subjects from two patient populations will be enrolled in order to test ultrasound technologies. A total of 30 subjects between 2-5 years of age will be enrolled.

1. 15 children with increased liver stiffness due to the Fontan operation
2. 15 children with increased liver stiffness caused by Biliary Atresia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 2-5 years
* Children who are scheduled to have a Stage 3 Fontan cardiac operation (arm 1) AND Children who have chronic liver disease caused by biliary atresia (arm 2)
* Patient must be receiving care at the University of Michigan CS Mott Children's Hospital
* Parent/guardian must be willing to sign the study consent form

Exclusion Criteria:

* For arm 1 subjects: pre-existing evidence of chronic liver disease (as defined by chronic elevation (over 4 weeks) of alanine aminotransferase (ALT), aspartate aminotransferase (AST), or conjugated bilirubin to greater than two times the upper limit of normal
* For arm 1 subjects: evidence of overt liver nodularity by conventional US imaging or evidence of portal vein or hepatic vein thrombosis (clots) by US Doppler exam

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients will either be scheduled for a Stage 3 Fontan cardiac operation or have chronic liver disease caused by biliary atresia.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Shear wave speed | 15 minutes
  Shear wave speed is a measure of stiffness of liver tissue expressed in units of m/s

CONTACTS AND LOCATIONS:
Overall Officials: Frank DiPaola, MD, Principal Investigator — University of Michigan
Locations (1):
- C.S. Mott Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No